CLINICAL TRIAL: NCT04693780
Title: Randomized Controlled Trial of Citizen-targeted Evidence-based Resources for Patients, Family Members and Caregivers Seeking Health Information
Brief Title: Randomized Controlled Trial of Citizen-targeted Evidence-based Resources
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, John Lavis, Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 8180
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Bowel Diseases; Irritable Bowel Syndrome
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Both the intervention and control groups will continue for three months. After three months, the control group will be sent a message highlighting some additions to the content provided to them. From his point forward when they login to the system they will be presented with the same content that was previously only available to the intervention group. Providing those in the control group access to the same material as the intervention group for a period of the study will allow for direct within- group comparison as well as a direct comparison between groups. Both groups will continue in this manner for an additional three months.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Once randomized, each participant will be allocated to their respective group by the website programmers who will allocate based on identification number and will not be privy to personal information regarding the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured guide with pre-appraisal content (Experimental): Once logged into the website, participants in the intervention group will navigate health information through an annotated structured guide to health evidence which is designed to inform participants where to find specific health information but it will also provide information to understand why such content is more valuable than other content. This structured annotated guide to evidence will also outline the value of pre-appraisal and will help them navigate to products produced for them. These products have been produced by the research team and include a collection of web resource ratings, evidence summaries and blog posts modelled after those developed and presented on the McMaster Optimal Aging Portal. The topics of this citizen content match the scope of the IMAGINE Network.
  Interventions: Other: Structured guide
- Listing without pre-appraisal content (Placebo Comparator): Once logged into the website, participants in the control group will navigate health information through a structured one-page guide (see Appendix 1) that does not include pre-appraisal information. Instead it will list the main organizations in the field that produce citizen content with descriptions of the type of content they produce with links to their individual websites. This will be presented to participants when they login to the platform. None of the citizen content produced specifically for the study will be provided to them prior to crossing-over.
  Interventions: Other: List

INTERVENTIONS:
Other: Structured guide — Structured guide
  Arms: Structured guide with pre-appraisal content
Other: List — List
  Arms: Listing without pre-appraisal content

SUMMARY:
The purpose of this study is to determine whether an online resource developed to aid health consumers in making health decisions and better support them to seek quality evidence before other evidence is effective in the context of inflammatory bowel disease and irritable bowel syndrome

DETAILED DESCRIPTION:
Participants who consent to participate in the study will be randomly allocated to either the intervention or control group.

Once logged into the website, participants in the intervention group will navigate health information through an annotated structured guide to health evidence (see Appendix 2) which is designed to inform participants where to find specific health information but it will also provide information to understand why such content is more valuable than other content. This structured annotated guide to evidence will also outline the value of pre-appraisal and will help them navigate to products produced for them. These products have been produced by the research team and include a collection of web resource ratings, evidence summaries and blog posts modelled after those developed and presented on the McMaster Optimal Aging Portal.

Once logged into the website, participants in the control group will navigate health information through a structured one-page guide (see Appendix 1) that does not include pre-appraisal information. Instead it will list the main organizations in the field that produce citizen content with descriptions of the type of content they produce with links to their individual websites. This will be presented to participants when they login to the platform. None of the citizen content produced specifically for the study will be provided to them prior to crossing-over.

All participants will receive periodic reminders to access the content in the form of an email sent every two weeks.

Both the intervention and control groups will continue for three months. After three months, the control group will be sent a message highlighting some additions to the content provided to them. From his point forward when they login to the system they will be presented with the same content that was previously only available to the intervention group. Providing those in the control group access to the same material as the intervention group for a period of the study will allow for direct within- group comparison as well as a direct comparison between groups. Both groups will continue in this manner for an additional three months.

ELIGIBILITY:
Inclusion Criteria:

* Patients, caregivers or family members
* Aged 18 and above
* Have lived experience with, and are seeking information about, any of inflammatory bowel disease (i.e. Crohn's disease and ulcerative colitis), or irritable bowel syndrome

The study may also include, but will not initial target/recruit, patients, caregivers or family members, aged 18 and above, who have lived experience with, and are seeking information about all other gastrointestinal conditions and their symptoms (including abdominal pain, bloating, constipation, cramping, diarrhea, fatigue, gas, loss of appetite, nausea, and stools with mucus), microbiome and metabolomics, and celiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Are you:
  1. male
  2. female
  3. I do not identify as male or female
Enrollment: 200 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Website logins | Three months
  The primary outcome of the study is number of logins to the website that contains the health information (each log-in will be tracked using Google Analytics)

SECONDARY OUTCOMES:
Self-reported change in information usage | Baseline, 3 months, and 6 months
  Change in behaviour in regards to information usage collected through a questionnaire
Clicks on resources | Three months before cross-over and three months after cross-over
  Clicks on resources included in the guide/list with data compiled through Google Analytics
Time on website | Three months before cross-over and three months after cross-over
  Time on website with data compiled through Google Analytics

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Health Forum Impact Lab, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No